CLINICAL TRIAL: NCT02366702
Title: Kinematic, Kinetic, and Metabolic Comparison of Bilateral Transfemoral Ambulation With Passive Versus Powered Prosthetic Devices
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Southern California Institute for Research and Education (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Dana Craig, Health System Specialist, Southern California Institute for Research and Education
Other Study IDs: 01329
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Amputation; Artificial Limbs; Energy Expenditure; Kinetics

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Individuals with Bilateral Transfemoral Amputation
  Interventions: Device: Lower Limb Powered Knee-Ankle Prosthesis

INTERVENTIONS:
Device: Lower Limb Powered Knee-Ankle Prosthesis

SUMMARY:
The purpose of this descriptive and exploratory pilot study is to investigate: (1) sagittal plane hip kinematics and kinetics and (2) metabolic consumption/cost, for bilateral transfemoral walking with passive prostheses versus powered prostheses. The pilot study will collect data from three subjects with bilateral transfemoral amputations. Differences in kinetics, kinematics, and oxygen consumption/cost when comparing passive and powered components may indicate benefits for clinical application of powered devices for persons with lower limb amputation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* All causes of limb amputation: congenital, trauma, vascular, limb salvage, infection.
* All transfemoral residual limb lengths: joint disarticulation, long, medium, short, very short.
* Subjects currently walk with entirely passive type prostheses daily.
* Subjects walk without assistive devices OR with single point cane.
* High-activity level walkers

Exclusion Criteria:

* Ages < 18 or > 45 years
* Medical comorbidities or existing conditions that may impede the subjects ability to complete the protocol excluding the amputations.
* Current medications or pharmaceutical interventions that may impede the subjects ability to complete the protocol.
* Any powered prosthetic component or prosthesis, including but not exclusive to: Ossur Proprio Foot, BiOM or BiOM T2 System Foot, Ossur Power Knee, Ossur Symbionic Leg.
* Subjects requiring a walker, crutches, quad cane, or other assistive devices excluding a single point cane.
* Low-activity level walkers

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals with bilateral transfemoral amputation who are community level ambulators. Individuals are ambulatory with non-powered prosthetic devices.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Sagittal Plane Hip Moment | During the stance phase of the gait cycle after two weeks of training with powered device.
Metabolic Cost of Transport | 5 minutes of steady state walking after two weeks of training with powered device.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldfarb, Ph.D., Principal Investigator — Vanderbilt University
Locations (1):
- VA Long Beach Healthcare System, Long Beach, California, United States

REFERENCES:
- [Background] Ziegler-Graham K, MacKenzie EJ, Ephraim PL, Travison TG, Brookmeyer R. Estimating the prevalence of limb loss in the United States: 2005 to 2050. Arch Phys Med Rehabil. 2008 Mar;89(3):422-9. doi: 10.1016/j.apmr.2007.11.005. PMID 18295618
- [Background] Adams PF, Hendershot GE, Marano MA; Centers for Disease Control and Prevention/National Center for Health Statistics. Current estimates from the National Health Interview Survey, 1996. Vital Health Stat 10. 1999 Oct;(200):1-203. PMID 15782448
- [Background] Feinglass J, Brown JL, LoSasso A, Sohn MW, Manheim LM, Shah SJ, Pearce WH. Rates of lower-extremity amputation and arterial reconstruction in the United States, 1979 to 1996. Am J Public Health. 1999 Aug;89(8):1222-7. doi: 10.2105/ajph.89.8.1222. PMID 10432910
- [Background] Dougherty PJ, McFarland LV, Smith DG, Reiber GE. Combat-incurred bilateral transfemoral limb loss: a comparison of the Vietnam War to the wars in Afghanistan and Iraq. J Trauma Acute Care Surg. 2012 Dec;73(6):1590-5. doi: 10.1097/TA.0b013e318265fe64. PMID 23032809
- [Background] Kurdibaylo SF. Obesity and metabolic disorders in adults with lower limb amputation. J Rehabil Res Dev. 1996 Oct;33(4):387-94. PMID 8895133
- [Background] Wu YJ, Chen SY, Lin MC, Lan C, Lai JS, Lien IN. Energy expenditure of wheeling and walking during prosthetic rehabilitation in a woman with bilateral transfemoral amputations. Arch Phys Med Rehabil. 2001 Feb;82(2):265-9. doi: 10.1053/apmr.2001.19019. PMID 11239324
- [Background] Su PF, Gard SA, Lipschutz RD, Kuiken TA. Gait characteristics of persons with bilateral transtibial amputations. J Rehabil Res Dev. 2007;44(4):491-501. doi: 10.1682/jrrd.2006.10.0135. PMID 18247246
- [Background] Martinez-Villalpando EC, Herr H. Agonist-antagonist active knee prosthesis: a preliminary study in level-ground walking. J Rehabil Res Dev. 2009;46(3):361-73. PMID 19675988
- [Background] Hoffman MD, Sheldahl LM, Buley KJ, Sandford PR. Physiological comparison of walking among bilateral above-knee amputee and able-bodied subjects, and a model to account for the differences in metabolic cost. Arch Phys Med Rehabil. 1997 Apr;78(4):385-92. doi: 10.1016/s0003-9993(97)90230-6. PMID 9111458
- [Background] Quintero HA, Farris RJ, Ha K, Goldfarb M. Preliminary assessment of the efficacy of supplementing knee extension capability in a lower limb exoskeleton with FES. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:3360-3. doi: 10.1109/EMBC.2012.6346685. PMID 23366646
- [Background] Lawson BE, Huff A, Goldfarb M. A preliminary investigation of powered prostheses for improved walking biomechanics in bilateral transfemoral amputees. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:4164-7. doi: 10.1109/EMBC.2012.6346884. PMID 23366845
- [Background] Highsmith, M. J., Kahle, J. T., Carey, S. L., Lura, D. J., Dubey, R. V., & Quillen, W. S. (2010). Kinetic differences using a power knee and C-Leg while sitting down and standing up: a case report. JPO: Journal of Prosthetics and Orthotics, 22(4), 237-243
- [Background] Wolf, E. J., & Pruziner, A. L. (2014). Use of a Powered Versus a Passive Prosthetic System for a Person with Bilateral Amputations during Level-Ground Walking. JPO: Journal of Prosthetics and Orthotics, 26(3), 166-170
- [Background] Wolf EJ, Everding VQ, Linberg AA, Czerniecki JM, Gambel JM. Comparison of the Power Knee and C-Leg during step-up and sit-to-stand tasks. Gait Posture. 2013 Jul;38(3):397-402. doi: 10.1016/j.gaitpost.2013.01.007. Epub 2013 Jan 30. PMID 23375018
- [Background] Barr AE, Siegel KL, Danoff JV, McGarvey CL 3rd, Tomasko A, Sable I, Stanhope SJ. Biomechanical comparison of the energy-storing capabilities of SACH and Carbon Copy II prosthetic feet during the stance phase of gait in a person with below-knee amputation. Phys Ther. 1992 May;72(5):344-54. doi: 10.1093/ptj/72.5.344. PMID 1631203
- [Background] Barth, D. G., Schumacher, L., & Thomas, S. S. (1992). Gait analysis and energy cost of below-knee amputees wearing six different prosthetic feet. JPO: Journal of Prosthetics and Orthotics, 4(2), 63-75
- [Background] Snyder RD, Powers CM, Fontaine C, Perry J. The effect of five prosthetic feet on the gait and loading of the sound limb in dysvascular below-knee amputees. J Rehabil Res Dev. 1995 Nov;32(4):309-15. PMID 8770795
- [Background] Versluys R, Beyl P, Van Damme M, Desomer A, Van Ham R, Lefeber D. Prosthetic feet: state-of-the-art review and the importance of mimicking human ankle-foot biomechanics. Disabil Rehabil Assist Technol. 2009 Mar;4(2):65-75. doi: 10.1080/17483100802715092. PMID 19253096
- [Background] Hitt, J. K., Sugar, T. G., Holgate, M., & Bellman, R. (2010). An active foot-ankle prosthesis with biomechanical energy regeneration. Journal of medical devices,4(1), 011003
- [Background] Delussu AS, Brunelli S, Paradisi F, Iosa M, Pellegrini R, Zenardi D, Traballesi M. Assessment of the effects of carbon fiber and bionic foot during overground and treadmill walking in transtibial amputees. Gait Posture. 2013 Sep;38(4):876-82. doi: 10.1016/j.gaitpost.2013.04.009. Epub 2013 May 21. PMID 23702342
- [Background] Ferris AE, Aldridge JM, Rabago CA, Wilken JM. Evaluation of a powered ankle-foot prosthetic system during walking. Arch Phys Med Rehabil. 2012 Nov;93(11):1911-8. doi: 10.1016/j.apmr.2012.06.009. Epub 2012 Jun 22. PMID 22732369
- [Background] Sup, F., Bohara, A., & Goldfarb, M. (2007, April). Design and control of a powered knee and ankle prosthesis. In Robotics and Automation, 2007 IEEE International Conference on (pp. 4134-4139). IEEE
- [Background] Sup F, Varol HA, Mitchell J, Withrow TJ, Goldfarb M. Self-Contained Powered Knee and Ankle Prosthesis: Initial Evaluation on a Transfemoral Amputee. IEEE Int Conf Rehabil Robot. 2009 Jun 23;2009:638-644. doi: 10.1109/ICORR.2009.5209625. PMID 20228944
- [Background] McNealy LL, Gard SA. Effect of prosthetic ankle units on the gait of persons with bilateral trans-femoral amputations. Prosthet Orthot Int. 2008 Mar;32(1):111-26. doi: 10.1080/02699200701847244. PMID 18330810
- [Background] Gao F, Zhang F, Huang H. Investigation of sit-to-stand and stand-to-sit in an above knee amputee. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:7340-3. doi: 10.1109/IEMBS.2011.6091712. PMID 22256034
- [Background] Schmalz T, Blumentritt S, Marx B. Biomechanical analysis of stair ambulation in lower limb amputees. Gait Posture. 2007 Feb;25(2):267-78. doi: 10.1016/j.gaitpost.2006.04.008. Epub 2006 May 24. PMID 16725325
- [Background] Vrieling AH, van Keeken HG, Schoppen T, Otten E, Halbertsma JP, Hof AL, Postema K. Uphill and downhill walking in unilateral lower limb amputees. Gait Posture. 2008 Aug;28(2):235-42. doi: 10.1016/j.gaitpost.2007.12.006. Epub 2008 Feb 1. PMID 18242995
- [Background] Perry, J., Burnfield, J. M., & Cabico, L. M. (2010). Gait analysis: Normal and pathological function. Thorofare, NJ: SLACK
- [Background] Wolf SI, Alimusaj M, Fradet L, Siegel J, Braatz F. Pressure characteristics at the stump/socket interface in transtibial amputees using an adaptive prosthetic foot. Clin Biomech (Bristol). 2009 Dec;24(10):860-5. doi: 10.1016/j.clinbiomech.2009.08.007. Epub 2009 Sep 9. PMID 19744755
- [Background] Fradet L, Alimusaj M, Braatz F, Wolf SI. Biomechanical analysis of ramp ambulation of transtibial amputees with an adaptive ankle foot system. Gait Posture. 2010 Jun;32(2):191-8. doi: 10.1016/j.gaitpost.2010.04.011. Epub 2010 May 8. PMID 20457526
- [Background] Alimusaj M, Fradet L, Braatz F, Gerner HJ, Wolf SI. Kinematics and kinetics with an adaptive ankle foot system during stair ambulation of transtibial amputees. Gait Posture. 2009 Oct;30(3):356-63. doi: 10.1016/j.gaitpost.2009.06.009. Epub 2009 Jul 17. PMID 19616436
- [Background] Miller WC, Deathe AB, Speechley M. Lower extremity prosthetic mobility: a comparison of 3 self-report scales. Arch Phys Med Rehabil. 2001 Oct;82(10):1432-40. doi: 10.1053/apmr.2001.25987. PMID 11588750
- [Background] Torburn L, Powers CM, Guiterrez R, Perry J. Energy expenditure during ambulation in dysvascular and traumatic below-knee amputees: a comparison of five prosthetic feet. J Rehabil Res Dev. 1995 May;32(2):111-9. PMID 7562650
- [Background] Schmalz T, Blumentritt S, Jarasch R. Energy expenditure and biomechanical characteristics of lower limb amputee gait: the influence of prosthetic alignment and different prosthetic components. Gait Posture. 2002 Dec;16(3):255-63. doi: 10.1016/s0966-6362(02)00008-5. PMID 12443950
- [Background] Nolan L, Lees A. The functional demands on the intact limb during walking for active trans-femoral and trans-tibial amputees. Prosthet Orthot Int. 2000 Aug;24(2):117-25. doi: 10.1080/03093640008726534. PMID 11061198
- [Background] Frossard L, Cheze L, Dumas R. Dynamic input to determine hip joint moments, power and work on the prosthetic limb of transfemoral amputees: ground reaction vs knee reaction. Prosthet Orthot Int. 2011 Jun;35(2):140-9. doi: 10.1177/0309364611409002. PMID 21697197
- [Background] Ayyappa, E. (1997). Normal human locomotion, part 1: Basic concepts and terminology. JPO: Journal of Prosthetics and Orthotics, 9(1), 10-17
- [Background] Ayyappa, E. (1997). Normal human locomotion, Part 2: Motion, ground-reaction force and muscle activity. JPO: Journal of Prosthetics and Orthotics, 9(2), 49-57
- [Background] Waters RL, Perry J, Antonelli D, Hislop H. Energy cost of walking of amputees: the influence of level of amputation. J Bone Joint Surg Am. 1976 Jan;58(1):42-6. PMID 1249111
- [Background] Hughes J, Jacobs N. Normal human locomotion. Prosthet Orthot Int. 1979 Apr;3(1):4-12. doi: 10.3109/03093647909164693. PMID 471705
- [Background] Kadaba MP, Ramakrishnan HK, Wootten ME. Measurement of lower extremity kinematics during level walking. J Orthop Res. 1990 May;8(3):383-92. doi: 10.1002/jor.1100080310. PMID 2324857
- [Background] Darter BJ, Wilken JM. Energetic consequences of using a prosthesis with adaptive ankle motion during slope walking in persons with a transtibial amputation. Prosthet Orthot Int. 2014 Feb;38(1):5-11. doi: 10.1177/0309364613481489. Epub 2013 Mar 22. PMID 23525888
- [Background] Biswas, D., Roy, S., Lenka, P. K., & Kumar, R. (2010). Energy Cost and Gait Efficiency of Below-Knee Amputee and Normal Subject with Similar Physical Parameters & Quality of Life: A Comparative Case Study. Online Journal of Health and Allied Sciences, 9(3)
- [Background] Mohanty RK, Lenka P, Equebal A, Kumar R. Comparison of energy cost in transtibial amputees using "prosthesis" and "crutches without prosthesis" for walking activities. Ann Phys Rehabil Med. 2012 May;55(4):252-62. doi: 10.1016/j.rehab.2012.02.006. Epub 2012 Apr 10. English, French. PMID 22534430
- [Background] Cutti, A. G., Raggi, M., Garofalo, P., Giovanardi, A., Filippi, M. V., & Davalli, A. (2008). The effects of the 'Power Knee'prosthesis on amputees metabolic cost of walking and symmetry of gait-Preliminary results. Gait & Posture, 28, S38
- [Background] Herr HM, Grabowski AM. Bionic ankle-foot prosthesis normalizes walking gait for persons with leg amputation. Proc Biol Sci. 2012 Feb 7;279(1728):457-64. doi: 10.1098/rspb.2011.1194. Epub 2011 Jul 13. PMID 21752817
- [Background] Chin T, Sawamura S, Shiba R. Effect of physical fitness on prosthetic ambulation in elderly amputees. Am J Phys Med Rehabil. 2006 Dec;85(12):992-6. doi: 10.1097/01.phm.0000247653.11780.0b. PMID 17117003
- [Background] A. Cunha, E. Caetano, P. Ribeiro, G. Müller (eds.) Proceedings of the 9th International Conference on Structural Dynamics, EURODYN 2014. Porto, Portugal, 30 June - 2 July 2014
- [Background] Brockway JM. Derivation of formulae used to calculate energy expenditure in man. Hum Nutr Clin Nutr. 1987 Nov;41(6):463-71. PMID 3429265
- [Background] Schneider K, Hart T, Zernicke RF, Setoguchi Y, Oppenheim W. Dynamics of below-knee child amputee gait: SACH foot versus Flex foot. J Biomech. 1993 Oct;26(10):1191-204. doi: 10.1016/0021-9290(93)90067-o. PMID 8253824
- [Background] Simon AM, Ingraham KA, Fey NP, Finucane SB, Lipschutz RD, Young AJ, Hargrove LJ. Configuring a powered knee and ankle prosthesis for transfemoral amputees within five specific ambulation modes. PLoS One. 2014 Jun 10;9(6):e99387. doi: 10.1371/journal.pone.0099387. eCollection 2014. PMID 24914674
- [Background] Lawson BE, Ruhe B, Shultz A, Goldfarb M. A powered prosthetic intervention for bilateral transfemoral amputees. IEEE Trans Biomed Eng. 2015 Apr;62(4):1042-50. doi: 10.1109/TBME.2014.2334616. Epub 2014 Jul 2. PMID 25014950